CLINICAL TRIAL: NCT04919343
Title: A Randomised Controlled Trial to Evaluate the Efficacy of BBC Education's Tiny Happy People Content in Supporting Infant Language Development.
Brief Title: Do Video Materials Help Parents to Support Infant Development?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sheffield (Other)
Collaborators: University of Liverpool (Other); University of Manchester (Other); University of Melbourne (Other)
Responsible Party: Principal Investigator, Danielle Matthews, Reader in Cognitive Development, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 165718
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Language Development
Keywords: Vocabulary; socioeconomic status; Parenting; language; parent-child interaction; self-efficacy; infancy
MeSH Terms: conditions — Language

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BBC Tiny Happy People intervention (Experimental): Parents will be sent links each month directing them to BBC Tiny Happy People content via SMS text message using the secure service FireText. This content will be aimed at supporting language development. Parents will be asked to watch the video content and incorporate it into their parenting practices. The intervention will start when infants are aged 4-9 months and conclude when they are 18 months with a follow up to 24 months where time permits.
  Interventions: Behavioral: BBC Education Tiny Happy People videos
- Physical health control (Active Comparator): Similar to the experimental condition, parents will be sent links each month via SMS text message using FireText. These links will direct them to publicly available web content with tips to promote the healthy development of their baby, focusing on things such as healthy eating, physical activities, and dental care. The intervention will start when infants are aged 4-9 months and conclude when they are 18 months with a follow up to 24 months where time permits
  Interventions: Behavioral: Physical health control intervention

INTERVENTIONS:
Behavioral: BBC Education Tiny Happy People videos — This intervention involves regular texting of BBC Education Tiny Happy People videos to parents
  Arms: BBC Tiny Happy People intervention
Behavioral: Physical health control intervention — This intervention involves regular texting of publicly available videos about supporting infant physical and dental health to parents
  Arms: Physical health control

SUMMARY:
The aim of this project is to assess whether video materials from the BBC Tiny Happy People (THP) campaign are effective in terms of improving the language skills of socioeconomically disadvantaged children before they start school. This project will also look at how useable the service is for parents in terms of acceptability, effects on self-efficacy and implementation of advice.

DETAILED DESCRIPTION:
The current study will evaluate BBC Education's Tiny Happy People initiative (https://www.bbc.co.uk/tiny-happy-people) which seeks to reduce the impact of social and economic disadvantage on children's language skills before they arrive at primary school. BBC Education have created videos for parents and other caregivers with information about child development, tips and activities as well as other content of interest. The aim of the evaluation is to find out how parents feel about the materials and whether the videos promote a) caregiver confidence at 12, 18 and 24 months, b) caregiver-infant interaction at 12, 18 and 24 months and c) child language at 18 and 24 months. The primary outcome is expressive vocabulary size at 17-18 months. Families with 4- to 9-month-old infants who would like to take part will be randomly allocated either to a language support group or a physical health active control group and sent short, age-appropriate advice videos by text message three times a month until their children are 18 months old (with follow up videos for children until the age of 2 years where possible given study time limits).

ELIGIBILITY:
Inclusion Criteria:

Families must:

* be raising their child as a monolingual English speaker (at least 80% of the language they hear in the home is English)
* have a postcode in deciles 1-5 of the Office of National Statistics Index of Multiple Deprivation
* have access to the internet and a device to watch videos (via smart phone)

Infants must:

* be full term
* have a healthy birthweight

Exclusion Criteria:

Neither caregivers nor infants must have any significant known physical, mental or learning disability

Ages: 4 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 435 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
18 month expressive vocabulary | 2 months. Parents will complete the report within 2 months of the infant turning 18 months old.
  Infant expressive vocabulary, assessed using the communicative development inventory (CDI) at 18 months

SECONDARY OUTCOMES:
Caregiver responsive behaviour at 12, 18 and 24 months | Measures will be collected within 2 months of the child turning 12, 18 and 24 months
  Parents willing and able to upload a 5-minute video of a play time with their child will have the option to do so. A researcher will code the video using the PaRRis rating scale.
Caregiver self-efficacy at 12, 18 and 24 months | Measures will be collected within 2 months of the child turning 12, 18 and 24 months
  Parents will be sent a self-efficacy questionnaire to complete in the format of a qualtrics survey, via SMS text message at each time point. Questions will focus on how parents feel about their parenting in general and supporting their child's language development and physical health.
24 month expressive vocabulary | 3 months. Parents will complete the report within 3 months of the infant turning 24 months old.
  Infant expressive vocabulary, assessed using the communicative development inventory (CDI) at 24 months

OTHER OUTCOMES:
Intervention uptake - number of video links that were clicked on | Clicking on a video link within one month of it being sent
  Parents will be sent regular text messages with links to videos with information about supporting child language or physical health. We will take % of links clicked as a fidelity measure. We will check whether parents were more likely to click though to these links in one condition or the other and run a Complier Average Causal Effect analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Matthews, PhD, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised Individual Participant Data will be archived using the Open Science Framework's repository. For those participants who give permission, video data will also be archived such that researchers who have signed a confidentiality agreement can access this data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available at the same time as publication, anticipated within 2 years of study completion. It will remain available for at least 10 years.

REFERENCES:
- See also: Website hosting content for parents in language intervention arm — https://www.bbc.co.uk/tiny-happy-people